CLINICAL TRIAL: NCT03776734
Title: Effects of Different Durations of Cold Application on Respiratory Function, Exercise Capacity and Muscle Performance
Brief Title: Effects of Cold Application on Exercise Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, İlker Yatar, Senior İnstructor, Eastern Mediterranean University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ETK00-2017-0296
Record Dates: First submitted 2018-11-09; First posted 2018-12-17 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Cryotherapy Effect
Keywords: precooling; exercise; pulmonary function; isokinetic; lactate
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cryotherapy application (Experimental): effect of cold application
  Interventions: Other: Cryotherapy application

INTERVENTIONS:
Other: Cryotherapy application — Effects of 5-10- 20 minutes cold application on quadriceps muscle

SUMMARY:
It is of utmost importance to determine the individual upper limits in the recommended exercises for increasing the level of physical activity and for developing the cardiovascular system. Cardiovascular exercise tests are used in determining the exercise capacity and performance. Cardiovascular exercise tests allow maximal and submaximal loadings to determine the person's body temperature, oxygen consumption, fatigue, interpretation of cardiac responses, and exercise capacity.

Thermal equilibrium is achieved by the activation or inhibition of autonomic and behavioral thermocouples in order to generate, dissipate or protect heat. These thermocouples act together and allow precise control of body temperature, which is arranged in a narrow range.

Under certain conditions, such as body temperature, systemic inflammation, extreme environmental conditions, and exercise performance, it falls outside this narrow range. Metabolic heat production is 15 to 20 times greater than resting during exercise. In exercise performed under hot ambient conditions, the rate of heat production will exceed the rate of heat loss and cause it to rise rapidly before reaching a plateau. The increase due to the exhalation of body heat initiates two autonomous thermodynamics for heat dissipation: sweating and cutaneous vasodilatation. Although both mechanisms help prevent exaggerated increase in body temperature, they cause stress for the cardiovascular system.

Exercise performance and level of physical activity are influenced by individual characteristics such as personality adjustment and mediocre adjustment. Adaptation is defined as adaptation under natural conditions. Robinson showed that the individual salt losses are higher in individuals who exercise in a hot environment and cannot adapt to the temperature, a decrease in both urine and sweat salt contents with temperature compliance. One research has shown that exercise performance is influenced by heat-induced muscle cramps and cardiovascular function disorders due to this significant increase in salt loss. An increase in body temperature caused by exercise can have a negative impact on exercise performance and may lead to the development of conditions associated with increased body temperature.

Although many studies in literature have shown positive effects of performance of pre-exercise cold exercise on performance, there is no consensus on the use of cold applications.

DETAILED DESCRIPTION:
In our study, changes that may arise from individual differences will be tried to be controlled using repetitive measurements in the same individuals. Evaluation results will be recorded without any cold application in order to determine the circumstances prior to the application. In the following weeks, doses to both Quadriceps muscles will be recorded immediately after cold application of 5 minutes, 10 minutes and 20 minutes. Each of the applications will be held on the same day of the week and at the same time in 4 consecutive weeks. Nutritional and fluid trains (such as stimulant substances, amount of coffee tea), ambient conditions (temperature and humidity) that may affect individual performance will be recorded. Keeping room conditions under control will benefit from air conditioning. Individuals will be informed about the equipment and test protocol to be used in the tests. A sufficient number of trials will be done before the test so that the participants are familiar with the equipment and test protocol. All assessments will be performed by the same physiotherapist.

Participant Evaluation:

* Body composition will be assessed by height, weight, body fat percentage and skin thickness measurements. (TANİTA and Skinfold measurements)
* Bruce protocol with the aim of determining the exercise capacity (Bruce protocol installed on the treadmill), fatigue (lactate measurement device), heart rate (Polar wireless heart rate index), blood pressure (manual sphygmomanometer), saturated oxygen level (pulse oximetry) and oxygen consumption (metabolic gas analyzer) measurements.
* Respiratory Function Test (Spirometer, FEV1, FVC, FEV1 / FVC, FEF (25-75), PEF, MVV) should be performed for evaluation of respiratory functions.
* Respiratory muscle strength will be assessed by in-mouth pressure measurements (MIP-MEP device) during inhalation and exhalation.
* The application area will be assessed by dual laser infrared non-contact superficial temperature measurement thermometer and general body temperature infrared in-ear thermometer.
* Assessment of muscle strength and muscular endurance will be assessed with an isokinetic dynamometer.

Application Program:

Keeping room conditions, temperature and humidity under control will benefit from air conditioning. Temperature and humidity percentage indicator will be used when room conditions are monitored. Cooled ice packs of gel will be used to cool the quadriceps muscles. The amount of heat of the gel packets, before and after application of the application area, will be recorded by measuring with an infrared non-contact thermometer.

ELIGIBILITY:
Inclusion Criteria:

* Male, healthy individuals between the ages of 18-25
* individuals without peripheral circulatory disturbances
* Individuals without chronic disease
* Individuals without orthopedic, neurological, cardiopulmonary disturbances that may prevent evaluation and measurement
* individuals who have not exercised regularly in the past six months

Exclusion Criteria:

* Individuals with sensory loss
* Individuals with cold hypersensitivity
* Drug users who may influence performance

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 45 (Estimated)
Dates: Start 2018-07-30 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity | Before and after of each cold application. Each application will be applied same day and time of the week. All the application and measurement will take total 4 weeks for each subject.
  Oxygen consumption on maximal exercise test (Bruce Protocol) will be assessed with mobile metabolic analyzer system as expended oxygen level per kilogram in one minute (ml/kg/min.) will be measured after cold application.

SECONDARY OUTCOMES:
Muscle strength | Before and after of each cold application. Each application will be applied same day and time of the week. All the application and measurement will take total 4 weeks for each subject.
  Concentric quadriceps muscle torque values will be measured with isokinetic dynamometer as Newton-meter with speed of 60 and 240 degrees in seconds
Muscle endurance | Before and after of each cold application. Each application will be applied same day and time of the week. All the application and measurement will take total 4 weeks for each subject.
  Quadriceps muscle endurance values will be measured with isokinetic dynamometer as endurance percentage(%) with speed of 240 degrees in seconds
Forced expiratory volume | Before and after of each cold application. Each application will be applied same day and time of the week. All the application and measurement will take total 4 weeks for each subject.
  Forced expiratory volume in one second as liter (FEV1) will be measured with spirometry test
Forced vital capacity | Before and after of each cold application. Each application will be applied same day and time of the week. All the application and measurement will take total 4 weeks for each subject.
  Forced vital capacity as liter (FVC) will be measured with spirometry test
Peak expiratory flow | Before and after of each cold application. Each application will be applied same day and time of the week. All the application and measurement will take total 4 weeks for each subject.
  Peak expiratory flow as liter in one second (PEF) will be measured with spirometry test
Forced expiratory flow | Before and after of each cold application. Each application will be applied same day and time of the week. All the application and measurement will take total 4 weeks for each subject.
  Forced expiratory flow as liter (FEF25-75%) will be measured with spirometry test
Maximal voluntary ventilation | Before and after of each cold application. Each application will be applied same day and time of the week. All the application and measurement will take total 4 weeks for each subject.
  Maximal voluntary ventilation as liter in one minute (MVV) will be measured with spirometry test
Maximal inspiration pressure | Before and after of each cold application. Each application will be applied same day and time of the week. All the application and measurement will take total 4 weeks for each subject.
  Maximal inspiration pressure (MIP) represented by centimeters of water pressure (cmH2O) and measured with a manometer.
Maximal expiration pressure | Before and after of each cold application. Each application will be applied same day and time of the week. All the application and measurement will take total 4 weeks for each subject.
  Maximal expiration pressure (MEP) represented by centimeters of water pressure (cmH2O) and measured with a manometer.
Fatigue | Before and after of each cold application. Each application will be applied same day and time of the week. All the application and measurement will take total 4 weeks for each subject.
  Lactate level will be measured before and after maximal test.

CONTACTS AND LOCATIONS:
Overall Officials: İLKER YATAR, MSc. PT, Principal Investigator — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided